CLINICAL TRIAL: NCT02429310
Title: Adjuvant Benefit of Neuromuscular Electrical Stimulation to Supervised Exercise in Patients With Intermittent Claudication
Brief Title: Adjuvant Benefit of NMES to Supervised Exercise in Patients With IC
Acronym: AdjIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14HH2042
Record Dates: First submitted 2015-04-15; First posted 2015-04-29 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Intermittent Claudication; Peripheral Vascular Disease; Lower Limb Arterial Disease
Keywords: Intermittent Claudication; IC; Peripheral Arterial Disease; Peripheral Vascular Disease; Peripheral Arterial Occlusive Disease; Lower Limb Arterial Disease; Supervised Exercise Therapy; Supervised Exercise Programme; Exercise Therapy
MeSH Terms: conditions — Intermittent Claudication; Peripheral Vascular Diseases; Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supervised Exercise Only (No Intervention): This is the cohort of patients with Intermittent Claudication that will receive standard care of a supervised exercise programme only.
- NMES + Supervised Exercise (Experimental): This cohort of patients with Intermittent Claudication will receive the standard care of supervised exercise plus the use of a Revitive IX neuromuscular electrical stimulation device (Intervention) as per the protocol. The adjunctive benefit of the latter intervention compared to standard treatment alone will then be assessed.
  Interventions: Device: Revitive IX

INTERVENTIONS:
Device: Revitive IX — This is a neuromuscular electrical stimulation device
  Arms: NMES + Supervised Exercise

SUMMARY:
This study will assess the adjuvant benefit of a neuromuscular electrical stimulation device to standard treatment of supervised exercise in patients suffering from symptoms and effects of lower limb Intermittent Claudication.

DETAILED DESCRIPTION:
The circulation of blood around the body is dependent on effective pumping of the heart. Patients with claudication experience pain or discomfort in their legs usually during activity such as walking, which goes away at rest. Claudication is a symptom of peripheral arterial disease (PAD). If left untreated, patients can develop arterial insufficiency which can lead to various complications such as swelling, painful legs, reduced healing of injuries and the loss of limbs in extreme conditions.

PAD can be defined as a narrowing of the arteries reducing blood flow. It is most commonly due to atherosclerosis, and has associations with heart disease, stroke, and diabetes. Its incidence is estimated at 7-14% in the general population, increasing with age to about 20% in the over-seventies. It is associated with effects on mobility, skin condition and quality of life. Symptoms include pain in the legs on walking (intermittent claudication), pain at rest (particularly at night), gangrene, and limb loss. Management of PAD is based on encouraging exercise, and modification of risk factors such as smoking, high blood pressure, high cholesterol and diabetes.

In patients with PAD, exercise tolerance is often limited. Severe symptoms and disease can be treated by procedures such as balloon angioplasty, stenting or surgical bypass, but these procedures have risks. There also remains a percentage of patients who are not suitable for revascularisation, and have few options besides amputation available to them.

Current NICE guidelines (NICE Clinical Guideline 147: Lower Limb Peripheral Arterial Disease:Diagnosis and Management guidance.nice.org.uk/cg147) advise a supervised exercise programme should be offered to all patients with IC as well as best medical therapy. Regular exercise has shown to significantly improve symptoms of IC in patients, but the effects of this benefit quickly revert upon inactivity.

Some trials have shown that increasing the blood flow in the legs over time using medical devices (intermittent pneumatic compression, muscle stimulators), in addition to maximal medical and surgical therapy, can increase claudication distance, absolute walking distance, decrease rest pain, and reduce amputation rates. In our unit it has become apparent that there are an increasing number of medical devices available for circulatory support, either for use as an inpatient, out-patient, or a member of the general public. The supporting evidence for these is variable in scientific and clinical content or relevance, and requires clinical trials to evaluate further.

The device being used in this study activates the pumping action of the leg muscles by providing neuromuscular electrical stimulation (NMES) to cause foot muscle contraction and relaxation. This squeezes blood back towards the heart, improving circulation.

The investigators wish to evaluate whether NMES using this device has the same beneficial effects in patients with claudication when used in conjunction with supervised exercise.

ELIGIBILITY:
Inclusion Criteria:

* Patients with intermittent claudication who have the following are eligible for the study:

  * All ethnic groups, male or female above the age of 18 years.
  * Diagnosis of intermittent claudication
  * Be of non-childbearing potential; OR using adequate contraception and have a negative urine pregnancy test result within 24 hours, if appropriate, before using the study device.
  * Blood pressure currently under moderate control (< 160/100mmHg)
  * No current foot ulceration

Exclusion Criteria:

* Patients meeting any of the following criteria are to be excluded:

  * Has an unstable condition (eg, psychiatric disorder, a recent history of substance abuse) or otherwise thought to be unreliable or incapable of complying with the study protocol.
  * Has renal failure
  * Has diabetes
  * Has an ankle-brachial pressure index (ABPI) >0.9
  * Has any metal implants
  * Pregnant
  * Has a cardiac pacemaker or defibrillator device
  * Has recent lower limb injury or lower back pain
  * Has current foot ulceration or other skin ulcers
  * Has foot deformities
  * Has any disorder that, in the opinion of the Investigator, might interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alun H Davies, MA FRCS DM, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London - Charing Cross Hospital, London, Hammersmith, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Babber A, Ravikumar R, Onida S, Lane TRA, Davies AH. Effect of footplate neuromuscular electrical stimulation on functional and quality-of-life parameters in patients with peripheral artery disease: pilot, and subsequent randomized clinical trial. Br J Surg. 2020 Mar;107(4):355-363. doi: 10.1002/bjs.11398. Epub 2020 Jan 7. PMID 31912491

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Supervised Exercise Only | NMES + Supervised Exercise
Started | 22 | 20
Completed | 20 | 17
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Population: This includes all patients that were recruited. As per the participant flow module, 2 patients were lost in Supervised Exercise Only group after baseline assessment and 3 were lost in the NMES + Supervised Exercise group after baseline assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Supervised Exercise Only | NMES + Supervised Exercise | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11) | 66 (8) | 67 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 16 | 15 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 22 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Initial Walking Distance Measured by Treadmill
Description: For the initial claudication distance measurement, a fixed load treadmill test will be carried out at 3.5 km/h with a 10% gradient. The initial claudication distance (ICD) is the distance walked until the onset of pain.
Time Frame: Change in baseline treadmill walking distance at 6 weeks (positive numbers indicate increase from baseline, negative numbers indicate decrease from baseline) - 6 week - baseline values.
Measure: Median (Inter-Quartile Range); unit: metres
Arm/Group | Supervised Exercise Only | NMES + Supervised Exercise
Number analyzed (Participants) | 20 | 17
metres | 65.60 [33.98 to 93.88] | 95.50 [81.40 to 155.3]

2. Primary Outcome: Absolute Walking Distance Measured by Treadmill
Description: For the absolute claudication distance measurement, a fixed load treadmill test will be carried out at 3.5 km/h with a 10% gradient. The absolute claudication distance (ACD) is the distance walked before the participant is forced to stop due to typical pain.
Time Frame: Change in baseline treadmill walking distance at 6 weeks (positive numbers indicate increase from baseline, negative numbers indicate decrease from baseline)
Measure: Median (Inter-Quartile Range); unit: metres
Arm/Group | Supervised Exercise Only | NMES + Supervised Exercise
Number analyzed (Participants) | 20 | 17
metres | 146.7 [70.53 to 214.3] | 167.4 [102.7 to 229.2]

3. Secondary Outcome: Femoral Haemodynamics Measured by Femoral Artery Duplex Ultrasonography
Description: Ultrasound assessment of blood flow dynamics in the femoral artery will be obtained at rest, and if randomised to the intervention group, whilst using the device.
Time Frame: Change in baseline femoral haemodynamics at 6 weeks - 6 weeks - baseline.
Reporting Status: Not Posted

4. Secondary Outcome: Laser Doppler Flow Measured by Optical Laser
Description: Optical laser flowmetry probes will be used to assess the superficial skin circulation and temperature.
Time Frame: Change in baseline flowmetry at 6 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Symptomatic Scores by Questionnaire
Description: Validated questionnaires including the Edinburgh Claudication Questionnaire and Intermittent Claudication Questionnaire will be obtained at baseline and week 6.
Time Frame: Change in baseline questionnaire scores at 6 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Quality of Life Scores Measured by Questionnaire
Description: Validated questionnaires including the Euro-Quol 5D and Short Form 36 will be measured at baseline and 6 weeks.
Time Frame: Change in baseline quality of life at 6 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Urine Metabolic Profile
Description: A urine sample will be collected at baseline and at 6 weeks. Mass spectroscopy and nuclear magnetic resonance spectroscopy analysis will be carried out.
Time Frame: Change of profile at baseline and at 6 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Serum Metabolic Profile
Description: A serum sample will be collected at baseline and at 6 weeks. Mass spectroscopy and nuclear magnetic resonance spectroscopy analysis will be carried out.
Time Frame: Change of profile at baseline and 6 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: through participant's study completion, 1 year 10 months
Arm/Group | Supervised Exercise Only | NMES + Supervised Exercise
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/17
Other Adverse Events (participants affected / at risk) | 0/20 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes